CLINICAL TRIAL: NCT03631355
Title: Reducing Hemarthrosis in Anterior Cruciate Ligament Reconstruction With BTB Autograft by the Administration of Intravenous Tranexamic Acid: A Double-Blind Randomized Control Study
Brief Title: Reducing Hemarthrosis in ACL Reconstruction With BTB Autograft by the Administration of Intravenous TXA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-00538
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Anterior Cruciate Ligament Reconstruction
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACL Reconstruction w/ BTB Autograft + IV TXA (Active Comparator): Patients receive a standard arthroscopic ACL reconstruction with a BTB autograft. In addition, these selected patients received two individual doses of intravenous TXA intra-operatively.
  Interventions: Drug: Tranexamic Acid
- ACL Reconstruction w/ BTB Autograft, no IV TXA (No Intervention): Patients receive a standard arthroscopic ACL reconstruction with a BTB autograft. In addition, these selected patients did not receive two individual doses of intravenous TXA intra-operatively. Only the consented surgery was performed.

INTERVENTIONS:
Drug: Tranexamic Acid — One gram of intravenous tranexamic acid will be administered before tourniquet inflation and 1 gram of IV TXA before closure of the incision.
  Arms: ACL Reconstruction w/ BTB Autograft + IV TXA

SUMMARY:
The purpose of the proposed study is to evaluate the effects of administering intravenous tranexamic acid (TXA) to patients undergoing anterior cruciate ligament (ACL) reconstruction with bone-patellar tendon-bone autograft to minimize hemarthrosis within the knee joint and post operative pain.

DETAILED DESCRIPTION:
The purpose of the proposed study is to evaluate the effects of administering intravenous tranexamic acid (TXA) to patients undergoing anterior cruciate ligament (ACL) reconstruction with bone-patellar tendon-bone autograft to minimize hemarthrosis within the knee joint and post operative pain. Patients received the standard arthroscopic ACL reconstruction with a BTB autograft and were randomized to either receiving or not receiving two individual doses of TXA intra-operatively or receive. The goal of the study is to determine and evaluate the effect of intra-operative TXA on post-operative hemarthrosis, pain reduction, and opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

-PATIENTS UNDERGOING AN ACL RECONSTRUCTION WITH BTB AUTOGRAFT

Exclusion Criteria:

* Legally incompetent or mentally impaired (e.g., minors, Alzheimer's subjects, dementia, etc.)
* Younger than 18 years of age
* Any patient considered a vulnerable subject
* Have bleeding or clotting disorder
* Preoperative anticoagulation therapy
* Abnormal coagulation profile
* Renal disorder or insufficiency
* Sickle cell disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Alaia, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ACL Reconstruction w/ BTB Autograft, no IV TXA: Received a standard ACL Reconstruction w/ BTB Autograft without IV Tranexamic Acid
Period: Overall Study
Arm/Group | ACL Reconstruction w/ BTB Autograft + IV TXA | ACL Reconstruction w/ BTB Autograft, no IV TXA
Started | 55 | 55
Completed | 54 | 53
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACL Reconstruction w/ BTB Autograft + IV TXA | ACL Reconstruction w/ BTB Autograft, no IV TXA | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (5.8) | 29.7 (8.5) | 29.1 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 30 | 35 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 26.8 (5.2) | 26.1 (5.2) | 26.4 (5.2)
Operative Knee (Right, Left) [Count of Participants; unit: Participants]
  Operative Knee (Right) | 34 | 29 | 63
  Operative Knee (Left) | 21 | 26 | 47
Meniscal Repair (Yes, No) [Count of Participants; unit: Participants]
  Meniscal Repair (Yes) | 15 | 14 | 29
  Meniscal Repair (No) | 40 | 41 | 81
Meniscectomy (Yes, No) [Count of Participants; unit: Participants]
  Meniscectomy (Yes) | 24 | 23 | 47
  Meniscectomy (No) | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: POST-OPERATIVE HEMARTHROSIS
Description: Measured by assessing the operative knee at the first post-operative visit for the need of joint aspiration.
Time Frame: Post-operative week 1
Population: The patients in each respective arm were evaluated for knee joint hemarthrosis and prompted joint aspiration because of pain or significant swelling.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | ACL Reconstruction w/ BTB Autograft + IV TXA | ACL Reconstruction w/ BTB Autograft, no IV TXA
Number analyzed (Participants) | 23 | 26
ml | 26.7 (23.1) | 37.3 (23.2)

2. Primary Outcome: POST-OPERATIVE Opioid Consumption
Description: Each patient's opioid consumption was measured by morphine milligram equivalents (MME).
Time Frame: Days 1-7
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | ACL Reconstruction w/ BTB Autograft + IV TXA | ACL Reconstruction w/ BTB Autograft, no IV TXA
Number analyzed (Participants) | 54 | 53
MME | 130.9 (90.9) | 113.9 (85.0)

3. Primary Outcome: POST-OPERATIVE Patient Reported Pain Score on the Visual Analog Scale (VAS)
Description: Pain severity, measured by the Visual Analog Scale (VAS): a scale of 1-10, with 1 being the least amount of pain and 10 being the most amount of pain.
Time Frame: Post-operative day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACL Reconstruction w/ BTB Autograft + IV TXA | ACL Reconstruction w/ BTB Autograft, no IV TXA
Number analyzed (Participants) | 54 | 53
score on a scale | 2.7 (1.9) | 3.2 (1.8)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | ACL Reconstruction w/ BTB Autograft + IV TXA | ACL Reconstruction w/ BTB Autograft, no IV TXA
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

LIMITATIONS AND CAVEATS:
Possibility of observer bias is present as we did not perform in-office aspirations in patients in whom we thought the hemarthroses were not clinically significant, as these procedures can be painful and confer some risk of infection. Despite the decision to aspirate being made clinically, post-study analysis revealed no difference in the rate each surgeon performed an aspiration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT03631355/Prot_SAP_ICF_000.pdf